CLINICAL TRIAL: NCT03519516
Title: Phase I Clinical Trial, to Evaluate the Safety and Tolerability of the Ophthalmic Solution PRO-174 Versus Sophixín Ofteno®, Elaborated by Laboratorios Sophia on the Ocular Surface of Ophthalmological and Clinically Healthy Subjects
Brief Title: Safety and Tolerability of the PRO-174 Versus Sophixín Ofteno®, on the Ocular Surface of Healthy Subjects
Acronym: PRO-174/I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOPH174-0816/I
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Conjunctivitis; Conjunctivitis, Bacterial
Keywords: ocular antibiotic; quinolone; levofloxacin; ophthalmic antibiotic; antibiotic in drops
MeSH Terms: conditions — Conjunctivitis; Conjunctivitis, Bacterial

STUDY DESIGN:
Intervention Model Description: Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The blinding will correspond to the research subject and the principal investigator. In addition, the statistical analysis will be carried out in a blinded manner for the partial and final analysis.
  The masking will be done using boxes in the primary packaging identical in the two groups. Blinding for the research subject and the researcher will be done by replacing the commercial labels in the case of the comparator in the bottles and the use of identical labels that contain the allocation number.
  Blinding may be opened in the following cases:
  1. Presence of a serious adverse event.
  2. Safety alarm due to the use of the drugs under study.
  3. In case the sponsor determines it for any reason of security or other reason that considers pertinent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-174 (Experimental): Active ingredient: Levofloxacin 0.5%
  o Dosage: 1 drop in both eyes, 8 times a day during the waking period
  Interventions: Drug: PRO-174
- Sophixín Ofteno® (Active Comparator): o Dosage: 1 drop in both eyes, 8 times a day during the waking period
  Interventions: Drug: Sophixín Ofteno®

INTERVENTIONS:
Drug: PRO-174 — Pharmaceutical form: ophthalmic solution
  * Prepared by: Laboratorios Sophia, S.A. of C.V.
  * Description of the solution: transparent solution, free of visible particles.
  * Description of container: sterile multi-dose bottle
  Other Names: PRO174; Levofloxacin Ophthalmic Solution
  Arms: PRO-174
Drug: Sophixín Ofteno® — * Active substance: Ciprofloxacin 0.3%
  * Pharmaceutical form: Ophthalmic solution
  * Prepared by: Laboratorios Sophia, S.A. of C.V.
  * Description of the solution: transparent solution, free of visible particles.
  * Description of container: sterile multi-dose bottle
  Other Names: Ciprofloxacin Ophthalmic solution
  Arms: Sophixín Ofteno®

SUMMARY:
Phase I clinical trial, to evaluate the safety and tolerability of the ophthalmic solution PRO-174 versus Sophixín Ofteno®, elaborated by Laboratorios Sophia, S.A. of C.V. on the ocular surface of ophthalmologically and clinically healthy subjects.

Goals:

To evaluate the safety and tolerability of the formulation PRO-174 manufactured by Laboratorios Sophia, S.A. of C.V. on the ocular surface of clinically healthy subjects.

Hypothesis:

The ophthalmic solution PRO-174 presents a safety and tolerability profile similar to the comparator in healthy subjects.

DETAILED DESCRIPTION:
Phase I clinical trial, to evaluate the safety and tolerability of the ophthalmic solution PRO-174 versus Sophixín Ofteno®, elaborated by Laboratorios Sophia, S.A. of C.V. on the ocular surface of ophthalmologically and clinically healthy subjects.

Goals:

Methodology:

Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.

Number of patients:

30 subjects, divided into 2 groups [15 subjects (30 eyes) exposed per group]

Test product, dose and route of administration, lot number:

* PRO-174. Levofloxacin 0.5% ophthalmic solution. Prepared by Laboratorios Sophia, S.A. of C.V., Zapopan, Jalisco, Mexico.
* Dosage: 1 drop every 2 hours during the waking period (8 daily applications), on day 1 and 2; continuing with 1 drop every 4 hours during the waking period (4 daily applications) from day 3 to 7. Both eyes.
* Route of administration: ophthalmic

Duration of treatment: 7 days

Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for the quantitative variables. The qualitative variables will be presented in frequencies and percentages. The statistical analysis will be carried out through the Mann-Whitney U test for the quantitative variables for the difference between the groups. The intra-group difference will be made with the Wilcoxon rank test. The difference between the qualitative variables will be analyzed by means of X2 (Chi2). An alpha ≤ 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Systemically and ophthalmologically healthy subjects evaluated during the clinical history.
* Age between 18 to 45 years.
* Both genders.
* Blood tests (complete blood count, blood chemistry of three elements and liver function tests) within normal parameters specified by the reference laboratory with a lower and upper margin of 10%.
* Vital signs within normal parameters. (Vital signs at rest: blood pressure ≤ 139/89 mmHg, heart rate 60 -100 beats per minute and respiratory rate of 12-24 breaths per minute).
* Visual capacity 20/30 or better, in both eyes.
* Intraocular pressure ≥11 and ≤ 21 mmHg.

Exclusion Criteria:

General criteria

* Subjects with a history of hypersensitivity to any of the components of the research products.
* Subject users of topical ophthalmic medications of any pharmacological group.
* Subject users of medication by any other route of administration.
* Pregnant or lactating women.
* Women of childbearing age, who do not ensure a hormonal contraceptive method or intrauterine device during the study period or without a history of bilateral tubal obstruction, oophorectomy or hysterectomy; as fertile age we understand women who have not had their menopause, defined as 12 months since the last menstruation in women over 40 years.
* Subjects with participation in clinical research studies 90 days prior to inclusion in the present study.
* Diagnosis of liver disease or elevation to three times the normal upper value of any of the following liver enzymes: aspartate transferase (AST), alanine transferase (ALT) or bilirubin.
* Inability to attend or answer the evaluations made in each of the visits.
* Positive smoking (specified as cigarette consumption regardless of amount and frequency)
* Positive alcoholism (specified as the consumption of alcoholic beverages, regardless of quantity and frequency, during the study intervention period).
* Contact lens users.
* An occlusive iridocorneal angle, defined as a trabecular mesh visible at less than 90 ° from the angular circumference to gonioscopy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Private Medical Offices, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Villegas P, Navarro-Sanchez AA, Sanchez-Rios A, Olvera-Montano O, Baiza-Duran LM. Reexamining Ophthalmic Drugs, Safety and Tolerability in Phase 1 Clinical Trials. Ther Clin Risk Manag. 2021 Oct 21;17:1123-1134. doi: 10.2147/TCRM.S331294. eCollection 2021. PMID 34707360

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-174: Active ingredient: Levofloxacin 0.5%
  o Dosage: 1 drop in both eyes, 8 times a day during the waking period
  PRO-174: Pharmaceutical form: ophthalmic solution
  * Prepared by: Laboratorios Sophia, S.A. of C.V.
  * Description of the solution: transparent solution, free of visible particles.
  * Description of container: sterile multi-dose bottle
- Sophixín Ofteno®: o Dosage: 1 drop in both eyes, 8 times a day during the waking period
  Sophixín Ofteno®: o Active substance: Ciprofloxacin 0.3%
  * Pharmaceutical form: Ophthalmic solution
  * Prepared by: Laboratorios Sophia, S.A. of C.V.
  * Description of the solution: transparent solution, free of visible particles.
  * Description of container: sterile multi-dose bottle
Period: Overall Study
Arm/Group | PRO-174 | Sophixín Ofteno®
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: ophthalmologically and clinically healthy
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-174 | Sophixín Ofteno® | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.67 (4.15) | 28.93 (9.38) | 26.3 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (EAS)
Description: primary security variable the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent.
Time Frame: during the 12 days of evaluation, including the safety call (day 12).
Population: the analysis of the population was by protocol
Measure: Number; unit: adverse events
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
adverse events | 11 | 10
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.749, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Ocular Burning (OB)
Description: primary tolerability variable
  Ocular burning is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: the analysis of the study population was by protocol
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
percentage of participants
  Normal | 86.7 | 57.1
  Very mild | 6.7 | 14.3
  mild | 6.7 | 28.6
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.041, Chi-squared

3. Secondary Outcome: Intraocular Pressure (IOP)
Description: the intraocular pressure will be evaluated by means of the Goldman applanation tonometry whose unit of measurement is millimeters of mercury (mmHg), it is a continuous variable and its normality range is between 11 - 21 mmHg
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: The study population was analyzed by protocol
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
mmHg | 12.53 (1.0) | 12.68 (1.7)
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.694, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Breakup Time (BUT)
Description: breakup time lacrimal film is a continuous variable that will be measured in seconds, evaluating the time it takes to break it, is done by direct counting and the normality range and mayor to 10 seconds.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: The study population was analyzed by protocol
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
seconds | 15.27 (2.7) | 15.79 (2.9)
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.495, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Eyes With Epithelial Defects (ED) by Grade
Description: The epithelial defects will be evaluated by means of two stains, green lysine and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: The study population was analyzed by protocol
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
eyes
  Green lissamine grade 1 | 2 | 0
  Green lissamine grade 0 | 28 | 28
  luorescein grade 1 | 3 | 0
  fluorescein grade 0 | 27 | 28
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.492, Chi-squared — statistical analysis between groups for final visit with green lissamine
Statistical Analysis 2: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.238, Chi-squared, Corrected — statistical analysis between groups for final visit with fluorescein

6. Secondary Outcome: Percentage of Eyes With Conjunctival Hyperemia (CH) by Grade
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as Normal / Very Light / Mild / Moderate / Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Mild, moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: The study population was analyzed by protocol
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
percentage of eyes
  normal | 96.7 | 92.9
  very mild | 3.3 | 0
  Mild | 0 | 0
  moderate | 0 | 7.1
  severo | 0 | 0
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.213, Chi-squared

7. Secondary Outcome: Number of Eyes With Foreign Body Sensation (FBS) by Grade
Description: Foreign body sensation is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: The study population was analyzed by protocol
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
eyes
  Absent | 30 | 28
  Very mild | 0 | 0
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0

8. Secondary Outcome: Number of Eyes With Ocular Pruritus (P) by Grade
Description: Ocular pruritus is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: The study population was analyzed by protocol grade 1
Measure: Number; unit: number of eyes with Ocular pruritus
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
number of eyes with Ocular pruritus
  Absent | 24 | 24
  Very mild | 4 | 2
  Mild | 2 | 2
  Moderate | 0 | 0
  Severe | 0 | 0
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — it is considered as noninferiority if there is no difference greater than twenty percent between both medications; p = 0.741, Chi-squared, Corrected

9. Secondary Outcome: Number of Eyes of Chemosis
Description: The chemosis will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Population: the statistical analysis of the sample was performed by protocol
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
eyes | 0 | 0

10. Secondary Outcome: Visual Capacity
Description: The visual capacity variable will be reported using as a unit of measure a fraction, this is taken from a visual test with the Snellen primer, it is a Nominal type variable. where the optimal vision is 20/20 and higher scores indicate worse visual acuity.
  Snellen Scale: 20/200, 20/100, 20/70, 20/50, 20/40, 20/30, 20/25, 20/20, 20/15, 20/12, 20/10
  only the denominator of the fraction of each case is reported and averaged per group.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 7)
Measure: Mean (Standard Deviation); unit: units on a scale (snellen)
Units Other Than Participants: eyes
Arm/Group | PRO-174 | Sophixín Ofteno®
Number analyzed (Participants) | 15 | 14
Number analyzed (eyes) | 30 | 28
units on a scale (snellen) | 20.6 (2.17) | 20 (0)
Statistical Analysis 1: Comparison: PRO-174 vs Sophixín Ofteno®; Test type: Non-Inferiority — The study drug is considered non-inferior with respect to the comparator if there are no differences above twenty percent; p = 0.110, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: the adverse events were evaluated for a period of 13 days, from the baseline visit (day one) until the safety call three days after the last application of the study medication (day 13). MedDRA (V. 20.1)
Arm/Group | PRO-174 | Sophixín Ofteno®
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-174 (N=15) | Sophixín Ofteno® (N=15)
ocular burning (Eye disorders) | 5 (5) | 7 (7)
itching in the eye (Eye disorders) | 3 (3) | 1 (1)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
conjunctival hyperemia (Eye disorders) | 1 (1) | 0 (0)
tearing (Eye disorders) | 0 (0) | 1 (1)
skin rash (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
only the sponsor has the decision to disseminate or publish the information obtained from the investigation and the PIs involved must submit a formal request to the sponsor if they are willing to disseminate or publish such information, they may only publish them if they have the written authorization of the sponsor (Laboratoios Sophia S.A. de C.V.).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT03519516/Prot_SAP_000.pdf